CLINICAL TRIAL: NCT01597583
Title: MobileMedMinder: A Networked Aide for Medication Compliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Limaging (Unknown)
Responsible Party: Principal Investigator, Stephen Gottlieb, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HP-00051021
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Use of MobileMedMinder (Experimental)
  Interventions: Behavioral: Use of MobileMedMinder
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Use of MobileMedMinder — Use of an intervention to remind patients to take their medications.
  Arms: Use of MobileMedMinder

SUMMARY:
The main aim of this study is to conduct a randomized control trial to compare MobileMedMinder, a mobile phone based medication reminder software product, with currently accepted and empirically supported methods for increasing medication compliance through reminders and tracking.

ELIGIBILITY:
Inclusion Criteria:

* Taking beta blockers, ACE or ARB, and hydralazine for treatment of HF.

Exclusion Criteria:

* Inability to understand informed consent
* Inability to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Compliance | 3 months
  Pill counts will be used to assess compliance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States